CLINICAL TRIAL: NCT04008043
Title: The Effect of Dexamethasone vs Vicodin in Reducing Post-operative Pain After Periodontal Surgery Among Patients at the Henry M. Goldman School of Dental Medicine Pilot Study
Brief Title: Pilot Study: Effect of Dexamethasone vs Vicodin in Reducing Post-operative Pain
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Inadequate resources to start the study at this site.
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-38061
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Oral Surgery
Keywords: Dexamethasone; Vicodin; Pain management
MeSH Terms: conditions — Agnosia | interventions — acetaminophen, hydrocodone drug combination; Dexamethasone; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexamethasone (Experimental): Participants in this arm will take a 6mg dexamethasone tablet the day before surgery, a 6 mg tablet the day of surgery, a 4mg tablet the day after surgery and a 2mg tablet the second day after surgery. Pain scores will be recorded the evening of the surgery, the day after the surgery and one week after the surgery.
  Interventions: Drug: Dexamethasone
- Vicodin (Active Comparator): Participants in this arm will take a vicodin tablet every 4-6 hrs as needed to a maximum of 8 tablets after surgery. Each tablet has 300 mg acetaminophen and 5 mg hydrocodone. Pain scores will be recorded the evening of the surgery, the day after the surgery and one week after the surgery.
  Interventions: Drug: Vicodin

INTERVENTIONS:
Drug: Vicodin — In addition to taking one tablet of vicodin for pain every 4-6 hours up to 8 tablets, pain scores will be recorded the evening of the surgery, the day after the surgery and one week after the surgery.
  Other Names: acetaminophen and hydrocodone
  Arms: Vicodin
Drug: Dexamethasone — In addition to taking one tablet of dexamethasone for pain beginning the day before surgery and on the day of surgery, pain scores will be recorded the evening of the surgery, the day after the surgery and one week after the surgery.
  Other Names: corticosteroid
  Arms: Dexamethasone

SUMMARY:
The main objective of the pilot study is to investigate the process that includes recruitment (to estimate the rate of enrollment), feasibility, protocol refinement, and willingness of the subject to be randomized. To provide a sample estimate of the population parameter which is the true value in the target population to be used in the planning of a larger confirmatory study.

Secondary objectives include:

To examine the efficacy of pre/post-operational administration of dexamethasone vs Vicodin (acetaminophen and hydrocodone) for post-operative pain control following periodontal surgery at the Henry M. Goldman School of Dental Medicine.

To examine how BMI alters the response to dexamethasone and hydrocodone following periodontal surgery since obese patients have shown higher pain scores and increased pain sensitivity in previous experimental models of pain.

ELIGIBILITY:
Inclusion Criteria:

* Must be scheduled for periodontal surgery
* Subjects must be aged 21 years old and above
* Able and willing to provide informed consent
* 20 non-obese patients with BMI less than 30kg/m2
* 20 obese patients with BMI greater than or equal to 30kg/m2
* Diabetic and hypertensive patients included

Exclusion Criteria:

* Patients allergic to any formulations used in the study
* Patients with chronic use of nonsteroidal anti-inflammatory drugs or chronic use of narcotics; chronic defined as frequent use or misuse/ abuse so much as once a month
* Pregnant or lactating female patients; pregnancy test will be performed alongside the medical history
* Patients with kidney dysfunction
* Patients at risk for infective endocarditis determined by the medical history or past medical records

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Study enrollment rate of eligible participants | 12 months
  The proportion of patients that provide consent for the study

SECONDARY OUTCOMES:
Number of participants with breakthrough pain | evening of the surgery, the day after the surgery and one week after the surgery
Number medications taken for breakthrough pain | evening of the surgery, the day after the surgery and one week after the surgery
Medications taken for breakthrough pain | evening of the surgery, the day after the surgery and one week after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Said, BDS, Principal Investigator — BU Goldman School of Dental Medicine
Locations (1):
- Henry M. Goldman School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No